CLINICAL TRIAL: NCT03400176
Title: Phase Ib Open-label Study of VAY736 and Ibrutinib in Patients With Chronic Lymphocytic Leukemia (CLL) on Ibrutinib Therapy
Brief Title: VAY736 in Combination With Ibrutinib in Patients With CLL on Ibrutinib
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Business reasons
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CVAY736Y2102; 5R01CA177292-09 (NIH)
Record Dates: First submitted 2018-01-09; First posted 2018-01-17 (Actual); Results first posted 2025-05-13 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Chronic Lymphocytic Leukemia (CLL)
Keywords: Ibrutinib; VAY736; Chronic lymphocytic leukemia; CLL; Bruton's Tyrosine Kinase; BTK mutation
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — ianalumab; ibrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose Escalation (Experimental): Increasing doses of VAY736 in combination with a fixed dose of ibrutinib.
  Interventions: Drug: VAY736; Drug: ibrutinib
- Dose expansion (Experimental): Evaluation of the MTD/RD of the combination of VAY736 and ibrutinib that was identified in dose escalation.
  Interventions: Drug: VAY736; Drug: ibrutinib

INTERVENTIONS:
Drug: VAY736 — Experimental
Drug: ibrutinib — Approved medication
  Other Names: Imbruvica

SUMMARY:
Patients enrolled to the study had chronic lymphocytic leukemia (CLL) and received ibrutinib. Patients had either received ibrutinib for one year without having had a complete response or patients developed a resistance mutation to ibrutinib. This study had two parts, a dose escalation part and a dose expansion part.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CLL per the WHO classification
* At least 18 years of age
* Lack of a complete response after receiving ibrutinib for > 1 year OR presence of known ibrutinib resistance mutation
* Actively receiving ibrutinib at either 420 mg (patients enrolled to the escalation arm) or at a stable dose for at least 2 months prior to starting study treatment (patients enrolled to the expansion arm)

Exclusion Criteria:

* Known history of HIV
* Active hepatitis B or C infection
* Receipt of attenuated vaccine within 2 weeks prior to starting study treatment.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2018-04-09 (Actual); Primary Completion 2023-09-29 (Actual); Study Completion 2023-09-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - University of California San Diego - Moores Cancer Center, La Jolla, California
  - David Geffen School of Medicine at UCLA, Los Angeles, California
  - Ohio ST Compr Cancer Ctr James Hosp, Columbus, Ohio
  - SCRI Oncology Partners, Nashville, Tennessee
  - Uni of Utah Huntsman Cancer Inst, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kipps TJ. Mining the Microenvironment for Therapeutic Targets in Chronic Lymphocytic Leukemia. Cancer J. 2021 Jul-Aug 01;27(4):306-313. doi: 10.1097/PPO.0000000000000536. PMID 34398557
- See also: A Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=2319

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 39 patients were enrolled in the study. Fifteen patients participated in the dose escalation part across four treatment arms: VAY736 0.3 mg/kg Q2W + ibrutinib 420 mg, VAY736 1 mg/kg Q2W + ibrutinib 420 mg, VAY736 3 mg/kg Q2W + ibrutinib 420 mg, and VAY735 9 mg/kg + ibrutinib 420 mg. The remaining 24 subjects were enrolled in the expansion part and were treated with VAY736 3 mg/kg Q2W in combination with ibrutinib 420 mg or 280 mg.
Pre-assignment Details: The screening period began once patients had signed the study informed consent. Screening evaluations had to be completed within 21 days prior to the first dose of study treatment with the exception of baseline tumor assessments that could be conducted within 28 days prior to the first dose of study treatment. After screening, the treatment period started on Cycle 1 Day 1.
Groups:
- VAY736 0.3mg/kg Q2W + Ibrutinib 420mg: VAY736 0.3 mg/kg i.v. once every 2 weeks in combination with ibrutinib 420 mg oral once daily
- VAY736 1mg/kg Q2W + Ibrutinib 420mg: VAY736 1 mg/kg i.v. once every 2 weeks in combination with ibrutinib 420 mg oral once daily
- VAY736 3mg/kg Q2W + Ibrutinib 280mg: VAY736 3 mg/kg i.v. once every 2 weeks in combination with ibrutinib 280 mg oral once daily
- VAY736 3mg/kg Q2W + Ibrutinib 420mg: VAY736 3 mg/kg i.v. once every 2 weeks in combination with ibrutinib 420 mg oral once daily
- VAY736 9mg/kg Q2W + Ibrutinib 420mg: VAY736 9 mg/kg i.v. once every 2 weeks in combination with ibrutinib 420 mg oral once daily
Period: Dose Escalation
Arm/Group | VAY736 0.3mg/kg Q2W + Ibrutinib 420mg | VAY736 1mg/kg Q2W + Ibrutinib 420mg | VAY736 3mg/kg Q2W + Ibrutinib 280mg | VAY736 3mg/kg Q2W + Ibrutinib 420mg | VAY736 9mg/kg Q2W + Ibrutinib 420mg
Started | 4 | 3 | 0 | 4 | 4
Completed | 3 | 2 | 0 | 4 | 2
Not Completed | 1 | 1 | 0 | 0 | 2
Not completed — Progressive disease | 1 | 1 | 0 | 0 | 1
Not completed — Patient decision | 0 | 0 | 0 | 0 | 1
Period: Dose Expansion
Arm/Group | VAY736 0.3mg/kg Q2W + Ibrutinib 420mg | VAY736 1mg/kg Q2W + Ibrutinib 420mg | VAY736 3mg/kg Q2W + Ibrutinib 280mg | VAY736 3mg/kg Q2W + Ibrutinib 420mg | VAY736 9mg/kg Q2W + Ibrutinib 420mg
Started | 0 | 0 | 1 | 23 | 0
Group A (Chronic lymphocytic leukemia (CLL) patients on ibrutinib for one or more than one year with residual disease but without clinical relapse) | 0 | 0 | 0 | 19 | 0
Group B (Chronic lymphocytic leukemia (CLL) patients on ibrutinib with acquired resistance mutations but without clinical relapse) | 0 | 0 | 1 | 4 | 0
Completed | 0 | 0 | 0 | 19 | 0
Not Completed | 0 | 0 | 1 | 4 | 0
Not completed — Patient decision | 0 | 0 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 1 | 0
Not completed — Progressive disease | 0 | 0 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set: All patients who received at least one dose of study treatment in the dose escalation or dose expansion part of the study. Patients were analyzed according to the study treatment received.
Groups:
- Total: Total of all reporting groups
Arm/Group | VAY736 0.3mg/kg Q2W + Ibrutinib 420mg | VAY736 1mg/kg Q2W + Ibrutinib 420mg | VAY736 3mg/kg Q2W + Ibrutinib 280mg | VAY736 3mg/kg Q2W + Ibrutinib 420mg | VAY736 9mg/kg Q2W + Ibrutinib 420mg | Total
Number analyzed (Participants) | 4 | 3 | 1 | 27 | 4 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.3 (6.02) | 61.0 (1.73) | 57.0 | 63.5 (10.36) | 65.0 (10.42) | 63.9 (9.50)
Age, Customized [Count of Participants; unit: Participants]
  18 - < 65 years | 1 | 3 | 1 | 12 | 2 | 19
  65 - < 85 years | 3 | 0 | 0 | 15 | 2 | 20
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 0 | 7 | 3 | 11
  Male | 4 | 2 | 1 | 20 | 1 | 28
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 4 | 2 | 1 | 26 | 3 | 36
  Black or African American | 0 | 1 | 0 | 0 | 1 | 2
  Missing | 0 | 0 | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose-Limiting Toxicities (DLTs) in Cycle 1 (Escalation Only)
Description: A dose-limiting toxicity (DLT) is defined as an adverse event or abnormal laboratory value of Common Terminology Criteria for Adverse Events (CTCAE) grade ≥ 3 assessed as unrelated to disease, disease progression, inter-current illness or concomitant medications that occurs within the first 28 days of treatment with the combination of VAY736 and ibrutinib and meets the criteria defined in the study protocol. Other clinically significant toxicities may be considered to be DLTs, even if not CTCAE grade 3 or higher.
Time Frame: 28 days
Population: All patients in the dose escalation part who received at least one dose of study treatment and who either met the minimum exposure criterion defined in the protocol and had sufficient safety evaluations, or experienced a DLT during the first 28 days of treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | VAY736 0.3mg/kg Q2W + Ibrutinib 420mg | VAY736 1mg/kg Q2W + Ibrutinib 420mg | VAY736 3mg/kg Q2W + Ibrutinib 420mg | VAY736 9mg/kg Q2W + Ibrutinib 420mg
Number analyzed (Participants) | 4 | 3 | 4 | 4
Participants | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: Number of participants with AEs (any AE regardless of seriousness) and SAEs, including changes from baseline in vital signs, electrocardiograms and laboratory results qualifying and reported as AEs.
  AE grades to characterize the severity of the AEs were based on the Common Terminology Criteria for Adverse Events (CTCAE) version 4.03. For CTCAE v4.03, Grade 1 = mild; Grade 2 = moderate; Grade 3 = severe; Grade 4 = life-threatening; Grade 5 = death related to AE.
  All patients were followed for a 30-day safety follow-up period subsequent to completion of VAY736 therapy. No new AEs or SAEs were collected beyond the 30-day safety follow-up or during the efficacy follow up period.
Time Frame: From first dose of study treatment up to 30 days after the last dose of VAY736, up to approximately 8.8 months
Population: All patients who received at least one dose of study treatment in the dose escalation or dose expansion part of the study. Patients were analyzed according to the study treatment received.
Measure: Count of Participants; unit: Participants
Arm/Group | VAY736 0.3mg/kg Q2W + Ibrutinib 420mg | VAY736 1mg/kg Q2W + Ibrutinib 420mg | VAY736 3mg/kg Q2W + Ibrutinib 280mg | VAY736 3mg/kg Q2W + Ibrutinib 420mg | VAY736 9mg/kg Q2W + Ibrutinib 420mg
Number analyzed (Participants) | 4 | 3 | 1 | 27 | 4
Participants
  AEs | 4 | 3 | 1 | 27 | 4
  Treatment-related AEs | 2 | 2 | 1 | 15 | 1
  AEs with grade >=3 | 1 | 2 | 1 | 12 | 0
  Treatment-related AEs with grade >=3 | 0 | 1 | 1 | 7 | 0
  SAEs | 0 | 1 | 0 | 1 | 0
  Treatment-related SAEs | 0 | 1 | 0 | 1 | 0
  Fatal SAEs | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Participants With Dose Reductions and Dose Interruptions of VAY736
Description: For patients who did not tolerate the protocol-specified dosing schedule of the study drugs, dose adjustments could be permitted in order to allow the patient to continue study treatment.
Time Frame: Up to 7.8 months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | VAY736 0.3mg/kg Q2W + Ibrutinib 420mg | VAY736 1mg/kg Q2W + Ibrutinib 420mg | VAY736 3mg/kg Q2W + Ibrutinib 280mg | VAY736 3mg/kg Q2W + Ibrutinib 420mg | VAY736 9mg/kg Q2W + Ibrutinib 420mg
Number analyzed (Participants) | 4 | 3 | 1 | 27 | 4
Participants
  At least one dose reduction or interruption | 0 | 1 | 0 | 5 | 0
  At least one dose reduction | 0 | 0 | 0 | 1 | 0
  At least one dose interruption | 0 | 1 | 0 | 5 | 0

4. Primary Outcome: Number of Participants With Dose Reductions and Dose Interruptions of Ibrutinib
Description: as for outcome 3
Time Frame: Up to 8.5 months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | VAY736 0.3mg/kg Q2W + Ibrutinib 420mg | VAY736 1mg/kg Q2W + Ibrutinib 420mg | VAY736 3mg/kg Q2W + Ibrutinib 280mg | VAY736 3mg/kg Q2W + Ibrutinib 420mg | VAY736 9mg/kg Q2W + Ibrutinib 420mg
Number analyzed (Participants) | 4 | 3 | 1 | 27 | 4
Participants
  At least one dose reduction or interruption | 0 | 1 | 0 | 10 | 0
  At least one dose reduction | 0 | 0 | 0 | 0 | 0
  At least one dose interruption | 0 | 1 | 0 | 10 | 0

5. Primary Outcome: Dose Intensity of VAY736
Description: Dose intensity of VAY736 was calculated as: Actual Cumulative dose (mg/kg) / (Duration of exposure in weeks/2)
Time Frame: Up to 7.8 months
Population: as for outcome 2
Measure: Median (Full Range); unit: mg/kg/2 weeks
Arm/Group | VAY736 0.3mg/kg Q2W + Ibrutinib 420mg | VAY736 1mg/kg Q2W + Ibrutinib 420mg | VAY736 3mg/kg Q2W + Ibrutinib 280mg | VAY736 3mg/kg Q2W + Ibrutinib 420mg | VAY736 9mg/kg Q2W + Ibrutinib 420mg
Number analyzed (Participants) | 4 | 3 | 1 | 27 | 4
mg/kg/2 weeks | 0.30 [0.3 to 0.3] | 0.98 [0.9 to 1.0] | 3.00 [3.0 to 3.0] | 3.00 [1.4 to 3.0] | 8.97 [8.9 to 9.0]

6. Primary Outcome: Dose Intensity of Ibrutinib
Description: Dose intensity of ibrutinib was calculated as: Actual Cumulative dose (mg) / (Duration of exposure in days)
Time Frame: Up to 8.5 months
Population: as for outcome 2
Measure: Median (Full Range); unit: mg/day
Arm/Group | VAY736 0.3mg/kg Q2W + Ibrutinib 420mg | VAY736 1mg/kg Q2W + Ibrutinib 420mg | VAY736 3mg/kg Q2W + Ibrutinib 280mg | VAY736 3mg/kg Q2W + Ibrutinib 420mg | VAY736 9mg/kg Q2W + Ibrutinib 420mg
Number analyzed (Participants) | 4 | 3 | 1 | 27 | 4
mg/day | 420.00 [420.0 to 420.0] | 420.00 [407.7 to 420.0] | 280.00 [280.0 to 280.0] | 420.00 [395.7 to 420.0] | 420.00 [420.0 to 420.0]

7. Secondary Outcome: CR or CRi Rate at C9 for Expansion Arm A and Arm B by Investigator Per IWCLL
Description: Percentage of participants with Complete Response (CR) or Complete Response with Incomplete Marrow Recovery (CRi) by investigator assessment per International Working Group - Chronic Lymphocytic Leukemia (IWCLL) response criteria.
Time Frame: Cycle 9 Day 1 (C9). The duration of each cycle was 28 days.
Population: All patients who received at least one dose of study treatment in the dose expansion part of the study.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Groups:
- VAY736 3mg/kg Q2W Arm A + Ibrutinib 420mg: VAY736 3 mg/kg in combination with ibrutinib 420 mg in Dose Expansion Arm A: chronic lymphocytic leukemia (CLL) patients on ibrutinib for one or more than one year with residual disease but without clinical relapse
- VAY736 3mg/kg Q2W Arm B + Ibrutinib 280mg: VAY736 3 mg/kg in combination with ibrutinib 280 mg in Dose Expansion Arm B: chronic lymphocytic leukemia (CLL) patients on ibrutinib with acquired resistance mutations but without clinical relapse
- VAY736 3mg/kg Q2W Arm B + Ibrutinib 420mg: VAY736 3 mg/kg in combination with ibrutinib 420 mg in Dose Expansion Arm B: chronic lymphocytic leukemia (CLL) patients on ibrutinib with acquired resistance mutations but without clinical relapse
- All Patients Expansion: All patients in dose expansion arm A and arm B
Arm/Group | VAY736 3mg/kg Q2W Arm A + Ibrutinib 420mg | VAY736 3mg/kg Q2W Arm B + Ibrutinib 280mg | VAY736 3mg/kg Q2W Arm B + Ibrutinib 420mg | All Patients Expansion
Number analyzed (Participants) | 19 | 1 | 4 | 24
percentage of participants | 47.4 [27.4 to 68.0] | 0 [0 to 95.0] | 0 [0 to 52.7] | 37.5 [21.2 to 56.3]

8. Secondary Outcome: Posterior Mean of CR or CRi Response Rate at C9 for Expansion Arm A and Arm B (Bayesian Analysis)
Description: The rate of CR/CRi at C9 was analyzed for each expansion arm using a Bayesian modeling approach.
  A minimally informative beta distribution was used as prior distribution with parameters a=0.25 and b=1. This assumed, a priori, that the response rate was 20%.
  Values estimated from the model at Cycle 9 are presented in the table. Posterior geometric mean for CR/CRi rate and 90% credible intervals in each group are presented.
Time Frame: Cycle 9 Day 1 (C9). The duration of each cycle was 28 days.
Population: All patients who received at least one dose of study treatment in the dose expansion part of the study.
Measure: Geometric Mean (90% Confidence Interval); unit: percentage of participants
Arm/Group | VAY736 3mg/kg Q2W Arm A + Ibrutinib 420mg | VAY736 3mg/kg Q2W Arm B + Ibrutinib 280mg | VAY736 3mg/kg Q2W Arm B + Ibrutinib 420mg | All Patients Expansion
Number analyzed (Participants) | 19 | 1 | 4 | 24
percentage of participants | 45.68 [28.1 to 63.7] | 11.11 [0 to 51.6] | 4.76 [0 to 23] | 36.63 [21.8 to 52.7]

9. Secondary Outcome: Posterior Probability That the True CR or CRi Response Rate at C9 for Expansion Arm A and Arm B Falls in Pre-defined Activity Intervals (Bayesian Analysis)
Description: The rate of CR/CRi at C9 was analyzed for each expansion arm using a Bayesian modeling approach.
  A minimally informative beta distribution was used as prior distribution with parameters a=0.25 and b=1. This assumed, a priori, that the response rate was 20%.
  Values estimated from the model at Cycle 9 are presented in the table. The posterior probability that the true CR/CRi rate falls in the activity intervals defined below is presented:
  * [0, 20%) - clinically not meaningful
  * [20%, 40%) - moderate clinical benefit
  * [40%, 100%] - superior clinical benefit
Time Frame: Cycle 9 Day 1 (C9). The duration of each cycle was 28 days.
Population: All patients who received at least one dose of study treatment in the dose expansion part of the study.
Measure: Number; unit: percentage of participants
Arm/Group | VAY736 3mg/kg Q2W Arm A + Ibrutinib 420mg | VAY736 3mg/kg Q2W Arm B + Ibrutinib 280mg | VAY736 3mg/kg Q2W Arm B + Ibrutinib 420mg | All Patients Expansion
Number analyzed (Participants) | 19 | 1 | 4 | 24
percentage of participants
  [0, 20%) - clinically not meaningful | 0.5 | 80.2 | 93.6 | 3
  [20%, 40%) - moderate clinical benefit | 30.4 | 11.3 | 5.3 | 61.8
  40%, 100%] - superior clinical benefit | 69.1 | 8.5 | 1.1 | 35.2

10. Secondary Outcome: Overall Response Rate (ORR) Assessed by Investigator Per IWCLL in the Dose Escalation Part
Description: Efficacy was based on local investigator assessment per International Working Group - Chronic Lymphocytic Leukemia (IWCLL) response criteria.
  ORR per IWCLL is defined as the percentage of participants with a best overall response of Complete Response (CR), Complete Response with Incomplete Marrow Recovery (CRi) or Partial Response (PR).
Time Frame: Up to approximately 2.5 years
Population: All patients who received at least one dose of study treatment in the dose escalation part of the study.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Groups:
- All Patients Escalation: All patients in dose escalation arms
Arm/Group | VAY736 0.3mg/kg Q2W + Ibrutinib 420mg | VAY736 1mg/kg Q2W + Ibrutinib 420mg | VAY736 3mg/kg Q2W + Ibrutinib 420mg | VAY736 9mg/kg Q2W + Ibrutinib 420mg | All Patients Escalation
Number analyzed (Participants) | 4 | 3 | 4 | 4 | 15
percentage of participants | 50.0 [9.8 to 90.2] | 0 [0 to 63.2] | 50.0 [9.8 to 90.2] | 50.0 [9.8 to 90.2] | 40.0 [19.1 to 64.0]

11. Secondary Outcome: Overall Response Rate (ORR) Assessed by Investigator Per IWCLL in the Dose Expansion Part
Description: as for outcome 10
Time Frame: Up to approximately 2.7 years
Population: All patients who received at least one dose of study treatment in the dose expansion part of the study.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | VAY736 3mg/kg Q2W Arm A + Ibrutinib 420mg | VAY736 3mg/kg Q2W Arm B + Ibrutinib 280mg | VAY736 3mg/kg Q2W Arm B + Ibrutinib 420mg | All Patients Expansion
Number analyzed (Participants) | 19 | 1 | 4 | 24
percentage of participants | 84.2 [64.1 to 95.6] | 0 [0 to 95.0] | 25.0 [1.3 to 75.1] | 70.8 [52.1 to 85.4]

12. Secondary Outcome: Time to Progression (TTP) in the Dose Escalation Part
Description: Efficacy was based on local investigator assessment per International Working Group - Chronic Lymphocytic Leukemia (IWCLL) response criteria.
  TTP is defined as the time from start of treatment to date of event which is defined as the first documented progression or death due to underlying cancer.
  If a patient had not had an event, TTP was censored at the date of the last adequate disease assessment.
  TTP was analyzed using Kaplan-Meier estimates.
Time Frame: Up to approximately 2.5 years
Population: All patients who received at least one dose of study treatment in the dose escalation part of the study.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | VAY736 0.3mg/kg Q2W + Ibrutinib 420mg | VAY736 1mg/kg Q2W + Ibrutinib 420mg | VAY736 3mg/kg Q2W + Ibrutinib 420mg | VAY736 9mg/kg Q2W + Ibrutinib 420mg | All Patients Escalation
Number analyzed (Participants) | 4 | 3 | 4 | 4 | 15
months | 23.3 [2.8 to NA] — Not estimable due to insufficient number of participants with events. | 8.3 [1.8 to NA] — Not estimable due to insufficient number of participants with events. | 24.2 [5.6 to NA] — Not estimable due to insufficient number of participants with events. | 19.4 [2.8 to NA] — Not estimable due to insufficient number of participants with events. | 19.4 [2.8 to 25.1]

13. Secondary Outcome: Time to Progression (TTP) in the Dose Expansion Part
Description: as for outcome 12
Time Frame: Up to approximately 2.7 years
Population: All patients who received at least one dose of study treatment in the dose expansion part of the study.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | VAY736 3mg/kg Q2W Arm A + Ibrutinib 420mg | VAY736 3mg/kg Q2W Arm B + Ibrutinib 280mg | VAY736 3mg/kg Q2W Arm B + Ibrutinib 420mg | All Patients Expansion
Number analyzed (Participants) | 19 | 1 | 4 | 24
months | NA [26.3 to NA] — Not estimable due to insufficient number of participants with events. | 2.3 [NA to NA] — Not estimable due to insufficient number of participants with events. | NA [NA to NA] — Not estimable due to insufficient number of participants with events. | NA [26.3 to NA] — Not estimable due to insufficient number of participants with events.

14. Secondary Outcome: Percentage of Participants With Clearance of Ibrutinib Resistance Mutation During Treatment (up to C9) for Expansion Arm B
Description: Clearance was defined as less than 1% mutation bearing alleles (BTKC481 and/or PLCγ2) during treatment.
  Negative mutation is defined as having clearance of the baseline ibrutinib resistance mutation during treatment (up to Cycle 9 (C9)).
Time Frame: Up to Cycle 9 Day 1. The duration of each cycle was 28 days.
Population: All patients in the dose expansion arm B who received at least one dose of study treatment.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Groups:
- All Patients Expansion Arm B: All patients in dose expansion arm B
Arm/Group | VAY736 3mg/kg Q2W Arm B + Ibrutinib 280mg | VAY736 3mg/kg Q2W Arm B + Ibrutinib 420mg | All Patients Expansion Arm B
Number analyzed (Participants) | 1 | 4 | 5
percentage of participants | 0 [0 to 95.0] | 0 [0 to 52.7] | 0 [0 to 45.1]

15. Secondary Outcome: Maximum Observed Serum Concentration (Cmax) of VAY736
Description: Pharmacokinetic (PK) parameters were calculated based on VAY736 serum concentrations by using non-compartmental methods. Cmax is defined as the maximum (peak) observed concentration following a dose.
Time Frame: Pre-infusion and 2, 6, 24, 72, 168 and 336 hours after end of infusion on Cycle 1 Day 1 and Cycle 3 Day 1. The duration of the infusion was approximately 2 hours. 1 cycle=28 days
Population: Patients in the pharmacokinetic analysis set (PAS) who had an available value for the outcome measure at each timepoint. PAS consists of all patients who received one of the planned treatments, provided at least one primary PK parameter and did not vomit within 8 hours after the dosing of ibrutinib. Patients were analyzed according to the study treatment received.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | VAY736 0.3mg/kg Q2W + Ibrutinib 420mg | VAY736 1mg/kg Q2W + Ibrutinib 420mg | VAY736 3mg/kg Q2W + Ibrutinib 280mg | VAY736 3mg/kg Q2W + Ibrutinib 420mg | VAY736 9mg/kg Q2W + Ibrutinib 420mg
Number analyzed (Participants) | 4 | 3 | 1 | 27 | 4
µg/mL
  Cycle 1: number analyzed (Participants) | 4 | 2 | 1 | 26 | 4
  Cycle 1 | 9.61 (23.0) | 15.8 (59.8) | 65.9 | 59.4 (15.8) | 178 (26.7)
  Cycle 3: number analyzed (Participants) | 3 | 2 | 0 | 27 | 4
  Cycle 3 | 11.2 (21.2) | 21.6 (38.8) |  | 72.5 (33.9) | 260 (13.3)

16. Secondary Outcome: Time to Reach Maximum Serum Concentration (Tmax) of VAY736
Description: PK parameters were calculated based on VAY736 serum concentrations by using non-compartmental methods. Tmax is defined as the time to reach maximum (peak) concentration following a dose. Actual recorded sampling times were considered for the calculations.
Time Frame: as for outcome 15
Population: as for outcome 15
Measure: Median (Full Range); unit: hours
Arm/Group | VAY736 0.3mg/kg Q2W + Ibrutinib 420mg | VAY736 1mg/kg Q2W + Ibrutinib 420mg | VAY736 3mg/kg Q2W + Ibrutinib 280mg | VAY736 3mg/kg Q2W + Ibrutinib 420mg | VAY736 9mg/kg Q2W + Ibrutinib 420mg
Number analyzed (Participants) | 4 | 3 | 1 | 27 | 4
hours
  Cycle 1: number analyzed (Participants) | 4 | 2 | 1 | 26 | 4
  Cycle 1 | 4.30 [2.40 to 6.00] | 3.90 [2.00 to 5.80] | 2.20 [2.20 to 2.20] | 4.70 [2.00 to 6.10] | 5.80 [2.20 to 6.00]
  Cycle 3: number analyzed (Participants) | 3 | 2 | 0 | 27 | 4
  Cycle 3 | 2.00 [2.00 to 2.10] | 2.20 [2.10 to 2.30] |  | 2.10 [2.00 to 22.70] | 2.15 [0.00 to 2.70]

17. Secondary Outcome: Area Under the Serum Concentration-time Curve From Time Zero to the Time of the Last Quantifiable Concentration (AUClast) of VAY736
Description: PK parameters were calculated based on VAY7736 serum concentrations by using non-compartmental methods. The linear trapezoidal method was used for AUClast calculation.
Time Frame: as for outcome 15
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*µg/mL
Arm/Group | VAY736 0.3mg/kg Q2W + Ibrutinib 420mg | VAY736 1mg/kg Q2W + Ibrutinib 420mg | VAY736 3mg/kg Q2W + Ibrutinib 280mg | VAY736 3mg/kg Q2W + Ibrutinib 420mg | VAY736 9mg/kg Q2W + Ibrutinib 420mg
Number analyzed (Participants) | 4 | 3 | 1 | 27 | 4
hr*µg/mL
  Cycle 1: number analyzed (Participants) | 4 | 2 | 1 | 26 | 4
  Cycle 1 | 46.0 (29.1) | 55.5 (46.0) | 217 | 256 (19.1) | 930 (25.0)
  Cycle 3: number analyzed (Participants) | 3 | 2 | 0 | 27 | 4
  Cycle 3 | 75.6 (31.7) | 166 (48.2) |  | 368 (55.2) | 1780 (18.1)

18. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Ibrutinib
Description: PK parameters were calculated based on ibrutinib plasma concentrations by using non-compartmental methods. Cmax is defined as the maximum (peak) observed concentration following a dose.
Time Frame: Pre-dose and 0.5, 2, 6 and 24 hours post-dose on Cycle 1 Day 1 and Cycle 1 Day 8. 1 cycle=28 days
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | VAY736 0.3mg/kg Q2W + Ibrutinib 420mg | VAY736 1mg/kg Q2W + Ibrutinib 420mg | VAY736 3mg/kg Q2W + Ibrutinib 280mg | VAY736 3mg/kg Q2W + Ibrutinib 420mg | VAY736 9mg/kg Q2W + Ibrutinib 420mg
Number analyzed (Participants) | 4 | 3 | 1 | 27 | 4
ng/mL
  Cycle 1 Day 1: number analyzed (Participants) | 3 | 3 | 1 | 21 | 4
  Cycle 1 Day 1 | 93.5 (120.6) | 123 (28.8) | 212 | 83.3 (146.9) | 104 (62.7)
  Cycle 1 Day 8: number analyzed (Participants) | 4 | 3 | 0 | 26 | 3
  Cycle 1 Day 8 | 94.9 (84.4) | 158 (53.0) |  | 62.2 (149.4) | 97.0 (54.1)

19. Secondary Outcome: Time to Reach Maximum Plasma Concentration (Tmax) of Ibrutinib
Description: PK parameters were calculated based on ibrutinib plasma concentrations by using non-compartmental methods. Tmax is defined as the time to reach maximum (peak) concentration following a dose. Actual recorded sampling times were considered for the calculations.
Time Frame: Pre-dose and 0.5, 2, 6 and 24 hours post-dose on Cycle 1 Day 1 and Cycle 1 Day 8. 1 cycle=28 days
Population: as for outcome 15
Measure: Median (Full Range); unit: hours
Arm/Group | VAY736 0.3mg/kg Q2W + Ibrutinib 420mg | VAY736 1mg/kg Q2W + Ibrutinib 420mg | VAY736 3mg/kg Q2W + Ibrutinib 280mg | VAY736 3mg/kg Q2W + Ibrutinib 420mg | VAY736 9mg/kg Q2W + Ibrutinib 420mg
Number analyzed (Participants) | 4 | 3 | 1 | 27 | 4
hours
  Cycle 1 Day 1: number analyzed (Participants) | 3 | 3 | 1 | 21 | 4
  Cycle 1 Day 1 | 2.10 [1.90 to 2.10] | 2.00 [2.00 to 2.10] | 2.30 [2.30 to 2.30] | 2.10 [0.60 to 6.80] | 2.00 [1.90 to 2.20]
  Cycle 1 Day 8: number analyzed (Participants) | 4 | 3 | 0 | 26 | 3
  Cycle 1 Day 8 | 2.00 [1.50 to 6.00] | 2.00 [1.90 to 2.10] |  | 2.00 [0.50 to 2.50] | 2.00 [1.90 to 2.00]

20. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to the Time of the Last Quantifiable Concentration (AUClast) of Ibrutinib
Description: PK parameters were calculated based on ibrutinib plasma concentrations by using non-compartmental methods. The linear trapezoidal method was used for AUClast calculation.
Time Frame: Pre-dose and 0.5, 2, 6 and 24 hours post-dose on Cycle 1 Day 1 and Cycle 1 Day 8. 1 cycle=28 days
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*ng/mL
Arm/Group | VAY736 0.3mg/kg Q2W + Ibrutinib 420mg | VAY736 1mg/kg Q2W + Ibrutinib 420mg | VAY736 3mg/kg Q2W + Ibrutinib 280mg | VAY736 3mg/kg Q2W + Ibrutinib 420mg | VAY736 9mg/kg Q2W + Ibrutinib 420mg
Number analyzed (Participants) | 4 | 3 | 1 | 27 | 4
hr*ng/mL
  Cycle 1 Day 1: number analyzed (Participants) | 3 | 3 | 1 | 21 | 4
  Cycle 1 Day 1 | 541 (145.3) | 938 (63.4) | 890 | 696 (98.5) | 634 (34.6)
  Cycle 1 Day 8: number analyzed (Participants) | 4 | 3 | 0 | 26 | 3
  Cycle 1 Day 8 | 338 (69.6) | 552 (41.8) |  | 226 (134.0) | 323 (54.7)

21. Secondary Outcome: Number of Participants With Anti-VAY736 Antibodies
Description: VAY736 immunogenicity was evaluated in serum samples. Anti-drug antibodies (ADA) status was defined as follows:
  * ADA-negative at baseline: baseline sample where assay is ADA negative
  * ADA-positive at baseline: baseline sample where assay is ADA positive
  * ADA-negative post-baseline: ADA-negative sample at baseline and at least 1 post-baseline sample, all of which are ADA-negative samples
  * Treatment-induced ADA-positive: ADA-negative sample at baseline and at least 1 treatment-induced ADA-positive sample
  * Treatment-boosted ADA-positive: ADA-positive sample at baseline and at least 1 treatment-boosted ADA-positive sample
  * ADA-inconclusive post-baseline: patient who does not qualify for any of the above definitions
Time Frame: Baseline (before first dose) and post-baseline (assessed throughout the VAY736 treatment, up to 7.8 months).
Population: Patients who received at least 1 dose of VAY736 and had a determinant baseline immunogenicity (IG) sample and at least 1 determinant post-baseline IG sample for assessing anti-VAY736 antibodies. Patients were analyzed according to the study treatment received.
Measure: Number; unit: participants
Arm/Group | VAY736 0.3mg/kg Q2W + Ibrutinib 420mg | VAY736 1mg/kg Q2W + Ibrutinib 420mg | VAY736 3mg/kg Q2W + Ibrutinib 280mg | VAY736 3mg/kg Q2W + Ibrutinib 420mg | VAY736 9mg/kg Q2W + Ibrutinib 420mg
Number analyzed (Participants) | 4 | 3 | 1 | 27 | 4
participants
  ADA-negative at baseline | 4 | 3 | 1 | 24 | 4
  ADA-positive at baseline | 0 | 0 | 0 | 3 | 0
  ADA-negative post-baseline: number analyzed (Participants) | 4 | 3 | 1 | 24 | 4
  ADA-negative post-baseline | 4 | 3 | 1 | 24 | 4
  ADA-inconclusive post-baseline: number analyzed (Participants) | 4 | 3 | 1 | 24 | 4
  ADA-inconclusive post-baseline | 0 | 0 | 0 | 0 | 0
  Treatment-induced ADA-positive: number analyzed (Participants) | 4 | 3 | 1 | 24 | 4
  Treatment-induced ADA-positive | 0 | 0 | 0 | 0 | 0
  Treatment-boosted ADA-positive: number analyzed (Participants) | 4 | 3 | 1 | 24 | 4
  Treatment-boosted ADA-positive | 0 | 0 | 0 | 0 | 0

22. Post Hoc Outcome: All-Collected Deaths
Description: On-treatment deaths were collected from first dose of study treatment to 30 days after the last dose of VAY736. Post-treatment deaths were collected from 31 days after last dose of VAY736 until end of study. All deaths refer to the sum of on-treatment and post-treatment deaths.
Time Frame: On-treatment deaths: up to approximately 8.8 months. Post-treatment deaths: up to approximately 2.7 years
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | VAY736 0.3mg/kg Q2W + Ibrutinib 420mg | VAY736 1mg/kg Q2W + Ibrutinib 420mg | VAY736 3mg/kg Q2W + Ibrutinib 280mg | VAY736 3mg/kg Q2W + Ibrutinib 420mg | VAY736 9mg/kg Q2W + Ibrutinib 420mg
Number analyzed (Participants) | 4 | 3 | 1 | 27 | 4
participants
  On-treatment deaths | 0 | 0 | 0 | 0 | 0
  Post-treatment deaths | 0 | 0 | 0 | 1 | 0
  All deaths | 0 | 0 | 0 | 1 | 0

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected on-treatment, from first dose of study treatment up to 30 days after the last dose of VAY736, up to approximately 8.8 months. No AEs were collected in the post-treatment period. Deaths were collected on-treatment, from first dose of study treatment to 30 days after the last dose of VAY736, up to approximately 8.8 months. Post-treatment deaths were collected from 31 days after last dose of VAY736 until end of study, up to approximately 2.7 years.
Description: Deaths in the post-treatment period are not considered Adverse Events (AEs). No AEs were collected in the post-treatment period.
  Safety was analyzed in the Safety set including all patients who received at least one dose of study treatment in the dose escalation or dose expansion part of the study. Patients were analyzed according to the study treatment received.
Groups:
- VAY736 0.3mg/kg Q2W + Ibrutinib 420mg; VAY736 1mg/kg Q2W + Ibrutinib 420mg; VAY736 3mg/kg Q2W + Ibrutinib 280mg; VAY736 3mg/kg Q2W + Ibrutinib 420mg; VAY736 9mg/kg Q2W + Ibrutinib 420mg; All patients_On-treatment: Safety data up to 30 days after the last dose of VAY736
- VAY736 0.3mg/kg Q2W + Ibrutinib 420mg_Post-treatment; VAY736 1mg/kg Q2W + Ibrutinib 420mg_Post-treatment; VAY736 3mg/kg Q2W + Ibrutinib 280mg_Post-treatment; VAY736 3mg/kg Q2W + Ibrutinib 420mg_Post-treatment; VAY736 9mg/kg Q2W + Ibrutinib 420mg_Post-treatment: Deaths collected in the post-treatment period (starting from Day 31 after last dose of VAY736). No AEs were collected during this period.
Arm/Group | VAY736 0.3mg/kg Q2W + Ibrutinib 420mg | VAY736 1mg/kg Q2W + Ibrutinib 420mg | VAY736 3mg/kg Q2W + Ibrutinib 280mg | VAY736 3mg/kg Q2W + Ibrutinib 420mg | VAY736 9mg/kg Q2W + Ibrutinib 420mg | All patients_On-treatment | VAY736 0.3mg/kg Q2W + Ibrutinib 420mg_Post-treatment | VAY736 1mg/kg Q2W + Ibrutinib 420mg_Post-treatment | VAY736 3mg/kg Q2W + Ibrutinib 280mg_Post-treatment | VAY736 3mg/kg Q2W + Ibrutinib 420mg_Post-treatment | VAY736 9mg/kg Q2W + Ibrutinib 420mg_Post-treatment
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/3 | 0/1 | 0/27 | 0/4 | 0/39 | 0/4 | 0/3 | 0/1 | 1/27 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4 | 2/3 | 0/1 | 2/27 | 0/4 | 4/39 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 4/4 | 3/3 | 1/1 | 27/27 | 4/4 | 39/39 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | VAY736 0.3mg/kg Q2W + Ibrutinib 420mg (N=4) | VAY736 1mg/kg Q2W + Ibrutinib 420mg (N=3) | VAY736 3mg/kg Q2W + Ibrutinib 280mg (N=1) | VAY736 3mg/kg Q2W + Ibrutinib 420mg (N=27) | VAY736 9mg/kg Q2W + Ibrutinib 420mg (N=4) | All patients_On-treatment (N=39) | VAY736 0.3mg/kg Q2W + Ibrutinib 420mg_Post-treatment (N=0) | VAY736 1mg/kg Q2W + Ibrutinib 420mg_Post-treatment (N=0) | VAY736 3mg/kg Q2W + Ibrutinib 280mg_Post-treatment (N=0) | VAY736 3mg/kg Q2W + Ibrutinib 420mg_Post-treatment (N=0) | VAY736 9mg/kg Q2W + Ibrutinib 420mg_Post-treatment (N=0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | NA | NA | NA | NA | NA
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 1 | NA | NA | NA | NA | NA
Escherichia sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA
Neutrophil count decreased (Investigations) | 0 | 1 | 0 | 1 | 0 | 2 | NA | NA | NA | NA | NA
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | VAY736 0.3mg/kg Q2W + Ibrutinib 420mg (N=4) | VAY736 1mg/kg Q2W + Ibrutinib 420mg (N=3) | VAY736 3mg/kg Q2W + Ibrutinib 280mg (N=1) | VAY736 3mg/kg Q2W + Ibrutinib 420mg (N=27) | VAY736 9mg/kg Q2W + Ibrutinib 420mg (N=4) | All patients_On-treatment (N=39) | VAY736 0.3mg/kg Q2W + Ibrutinib 420mg_Post-treatment (N=0) | VAY736 1mg/kg Q2W + Ibrutinib 420mg_Post-treatment (N=0) | VAY736 3mg/kg Q2W + Ibrutinib 280mg_Post-treatment (N=0) | VAY736 3mg/kg Q2W + Ibrutinib 420mg_Post-treatment (N=0) | VAY736 9mg/kg Q2W + Ibrutinib 420mg_Post-treatment (N=0)
Anaemia (Blood and lymphatic system disorders) | 2 | 3 | 0 | 8 | 1 | 14 | NA | NA | NA | NA | NA
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA
Lymph node pain (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1 | 0 | 2 | NA | NA | NA | NA | NA
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 1 | NA | NA | NA | NA | NA
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA
Palpitations (Cardiac disorders) | 0 | 1 | 0 | 4 | 0 | 5 | NA | NA | NA | NA | NA
Sinus bradycardia (Cardiac disorders) | 1 | 0 | 0 | 1 | 0 | 2 | NA | NA | NA | NA | NA
Sinus tachycardia (Cardiac disorders) | 0 | 1 | 0 | 2 | 1 | 4 | NA | NA | NA | NA | NA
Cataract (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA
Retinal tear (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA
Vision blurred (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA
Vitreous floaters (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 3 | 0 | 4 | NA | NA | NA | NA | NA
Diarrhoea (Gastrointestinal disorders) | 0 | 3 | 0 | 2 | 2 | 7 | NA | NA | NA | NA | NA
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 3 | 0 | 4 | NA | NA | NA | NA | NA
Frequent bowel movements (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 4 | 1 | 6 | NA | NA | NA | NA | NA
Oral pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 4 | 0 | 5 | NA | NA | NA | NA | NA
Vomiting (Gastrointestinal disorders) | 0 | 2 | 0 | 2 | 0 | 4 | NA | NA | NA | NA | NA
Chills (General disorders) | 0 | 2 | 0 | 1 | 0 | 3 | NA | NA | NA | NA | NA
Fatigue (General disorders) | 0 | 1 | 0 | 7 | 0 | 8 | NA | NA | NA | NA | NA
Influenza like illness (General disorders) | 0 | 0 | 0 | 2 | 1 | 3 | NA | NA | NA | NA | NA
Malaise (General disorders) | 1 | 0 | 0 | 1 | 0 | 2 | NA | NA | NA | NA | NA
Non-cardiac chest pain (General disorders) | 0 | 1 | 0 | 1 | 0 | 2 | NA | NA | NA | NA | NA
Oedema peripheral (General disorders) | 0 | 1 | 0 | 2 | 0 | 3 | NA | NA | NA | NA | NA
Pyrexia (General disorders) | 0 | 2 | 0 | 0 | 0 | 2 | NA | NA | NA | NA | NA
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 2 | NA | NA | NA | NA | NA
Cystitis (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 2 | NA | NA | NA | NA | NA
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 2 | NA | NA | NA | NA | NA
Onychomycosis (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 2 | NA | NA | NA | NA | NA
Paronychia (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 2 | NA | NA | NA | NA | NA
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 2 | 1 | 3 | NA | NA | NA | NA | NA
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 2 | 2 | 5 | NA | NA | NA | NA | NA
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 2 | 1 | 3 | NA | NA | NA | NA | NA
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 1 | 3 | NA | NA | NA | NA | NA
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 3 | 0 | 3 | NA | NA | NA | NA | NA
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 0 | 2 | NA | NA | NA | NA | NA
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0 | 2 | NA | NA | NA | NA | NA
Vaccination complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 0 | 2 | NA | NA | NA | NA | NA
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 0 | 0 | 1 | 1 | NA | NA | NA | NA | NA
Alanine aminotransferase increased (Investigations) | 1 | 1 | 0 | 3 | 0 | 5 | NA | NA | NA | NA | NA
Amylase increased (Investigations) | 0 | 0 | 0 | 4 | 1 | 5 | NA | NA | NA | NA | NA
Aspartate aminotransferase increased (Investigations) | 1 | 1 | 0 | 3 | 0 | 5 | NA | NA | NA | NA | NA
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 0 | 2 | 0 | 3 | NA | NA | NA | NA | NA
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 4 | 0 | 4 | NA | NA | NA | NA | NA
Blood creatinine increased (Investigations) | 1 | 0 | 0 | 4 | 1 | 6 | NA | NA | NA | NA | NA
Blood iron decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 3 | 0 | 3 | NA | NA | NA | NA | NA
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 2 | 0 | 2 | NA | NA | NA | NA | NA
Lipase increased (Investigations) | 0 | 0 | 0 | 6 | 0 | 6 | NA | NA | NA | NA | NA
Lymphocyte count decreased (Investigations) | 2 | 0 | 0 | 6 | 0 | 8 | NA | NA | NA | NA | NA
Lymphocyte count increased (Investigations) | 2 | 1 | 0 | 2 | 0 | 5 | NA | NA | NA | NA | NA
Neutrophil count decreased (Investigations) | 1 | 3 | 0 | 4 | 1 | 9 | NA | NA | NA | NA | NA
Platelet count decreased (Investigations) | 1 | 2 | 0 | 2 | 0 | 5 | NA | NA | NA | NA | NA
Weight increased (Investigations) | 0 | 0 | 0 | 2 | 0 | 2 | NA | NA | NA | NA | NA
White blood cell count decreased (Investigations) | 1 | 2 | 0 | 2 | 0 | 5 | NA | NA | NA | NA | NA
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 3 | 0 | 10 | 1 | 16 | NA | NA | NA | NA | NA
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA
Hypernatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 2 | 2 | 0 | 7 | 1 | 12 | NA | NA | NA | NA | NA
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 7 | 0 | 9 | NA | NA | NA | NA | NA
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 0 | 2 | NA | NA | NA | NA | NA
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 1 | 3 | NA | NA | NA | NA | NA
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0 | 2 | NA | NA | NA | NA | NA
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 0 | 2 | NA | NA | NA | NA | NA
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 6 | 0 | 7 | NA | NA | NA | NA | NA
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 2 | 0 | 2 | 0 | 6 | NA | NA | NA | NA | NA
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 4 | 1 | 5 | NA | NA | NA | NA | NA
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 1 | 3 | NA | NA | NA | NA | NA
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 1 | 0 | 3 | NA | NA | NA | NA | NA
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 2 | 3 | NA | NA | NA | NA | NA
Osteoporosis postmenopausal (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | NA | NA | NA | NA | NA
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 5 | 1 | 6 | NA | NA | NA | NA | NA
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 2 | 0 | 2 | NA | NA | NA | NA | NA
Headache (Nervous system disorders) | 1 | 2 | 0 | 3 | 1 | 7 | NA | NA | NA | NA | NA
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 2 | 0 | 2 | NA | NA | NA | NA | NA
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 1 | NA | NA | NA | NA | NA
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA
Haematuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 1 | 2 | NA | NA | NA | NA | NA
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0 | 1 | 0 | 2 | NA | NA | NA | NA | NA
Renal colic (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 1 | NA | NA | NA | NA | NA
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 1 | NA | NA | NA | NA | NA
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 2 | 1 | 6 | NA | NA | NA | NA | NA
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 2 | 0 | 3 | NA | NA | NA | NA | NA
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1 | 0 | 3 | NA | NA | NA | NA | NA
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 1 | 3 | NA | NA | NA | NA | NA
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 2 | NA | NA | NA | NA | NA
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 0 | 2 | NA | NA | NA | NA | NA
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 2 | NA | NA | NA | NA | NA
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA
Hypertension (Vascular disorders) | 1 | 2 | 0 | 6 | 0 | 9 | NA | NA | NA | NA | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. Novartis does not prohibit any investigator from publishing. Any publications from a single site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2021-10-20): https://cdn.clinicaltrials.gov/large-docs/76/NCT03400176/Prot_000.pdf
  • Statistical Analysis Plan (2024-02-27): https://cdn.clinicaltrials.gov/large-docs/76/NCT03400176/SAP_001.pdf